CLINICAL TRIAL: NCT02519517
Title: Acute Permissive Hypercapnia During One Lung Ventilation: Impact on Right Ventricular Systolic and Diastolic Functions During Lung Resection
Brief Title: Permissive Hypercapnia During One Lung Ventilation: Impact on Right Ventricular Systolic and Diastolic Functions During Lung Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Hosny, Assistant (associate) professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: acute permissive hypercapnia
Record Dates: First submitted 2015-06-20; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- permissive hypercapnia (Experimental): during one lung ventilation, right ventricular function was assessed by TEE and the effect of rising PCO2 appreciated
  Interventions: Procedure: Permissive hypercapnia

INTERVENTIONS:
Procedure: Permissive hypercapnia — During one lung ventilation, right ventricular function was assessed by transesophageal echocardiography (TEE) and the effect of increased carbon dioxide pressure was evaluated

SUMMARY:
Investigators studied 15 patients scheduled for pulmonary resection through thoracotomy. Initial tidal volume (VT) 10ml kg-1 was reduced to 8ml kg-1 after one lung ventilation (OLV) and the rate adjusted to maintain partial pressure of arterial carbon dioxide (PaCO2) 30-35 mm Hg. Data were obtained at: T1, 15 min post establishing OLV with normocapnia, T2, 15 min post establishing OLV with hypercapnia (PaCO2 7.98kPa (60mmHg) and 9.31kPa (70mmHg) and pH >7.1), and T3, 15 min after resuming OLV with normocapnia. One-way repeated measures analysis of variance (ANOVA), with post hoc Dunnet´s test were used for analysis. A P value < 0.05 is considered statistically significant.

DETAILED DESCRIPTION:
Investigators studied 15 patients scheduled for elective pulmonary resection through thoracotomy. Patients had a standardized management for thoracotomies. Initial VT 10ml/ kg was reduced to 8ml/kg after OLV and the rate adjusted to maintain PaCO2 30-35 mm Hg. Haemodynamic, respiratory variables and echocardiographic data (Tei index and TAPSE) were obtained at: T1, 15 min post establishing OLV with normocapnia, T2, 15 min post establishing OLV with hypercapnia (PaCO2 7.98kPa (60mmHg) and 9.31kPa (70mmHg) and pH >7.1), and T3, 15 min after resuming OLV with normocapnia. One-way repeated measures ANOVA, with post hoc Dunnet´s test were used for analysis. A P value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* adult >18 yr
* elective pulmonary resection through thoracotomy.

Exclusion Criteria:

* Patients with pulmonary hypertension (systolic >50mmHg),
* intracranial hypertension or previous intracranial haemorrhage,
* pre-existing hypercapnia,
* co-existing metabolic acidosis,
* ischaemic heart disease,
* predicted postoperative FEV1<800 ml or <40% of the expected in pneumonectomy
* patient in which transesophageal echocardiography was contraindicated or necessary measurements were difficult to assess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Right ventricular systolic and diastolic functions measured by Tei index | Intraoperative
  Tei index and Tricuspid Annular Plane Systolic Excursion (TAPSE) were used to assess both RV systolic and diastolic functions